

IIS-F-PG-22-02 Edición: 4.2 Página 1 de 18

| A cumplimentar por el IIS La Fe | Nº referencia: |
|---------------------------------|-------------------|
| | Fecha de entrada: |

Una vez aprobado este proyecto su duración será de <u>5 años.</u> Transcurrido dicho periodo, sí considera que el proyecto no ha finalizado, deberá solicitar la ampliación del plazo de ejecución.

**Título del proyecto**<sup>1</sup>: Desarrollo de una crema protectora frente a las radiodermitis causadas por la radioterapia.

Acrónimo: RADIOCREMVAL

## Datos del Investigador/ a principal:

Nombre y apellidos: Antonio J. Conde Moreno

Servicio: Oncología Radioterápica

Valencia a 24 de enero de 2023

Antonio J. Conde Moreno Firma Investigador/a Principal

 $<sup>^{1</sup>_1}$ Modelo para presentar proyectos de Investigación básica-clínica (no equiparables a ensayos clínicos), por iniciativa de los grupos de investigación del IIS La Fe



#### Memoria de solicitud: Proyecto de investigación propio

IIS-F-PG-22-02 Edición: 04 Página 2 de 18

#### RESUMEN EJECUTIVO DEL PROYECTO

(máximo 500 palabras, antecedentes / justificación, hipótesis/objetivos y metodología):

La crema de estudio se va a evaluar en un estudio clínico controlado, aleatorio y multicentro realizado en 2 Hospitales, en el servicio de Oncología Radioterápica de Valencia para evaluar su efecto radioprotector y radiomitigador en el tratamiento profiláctico de la radiodermitis aguda por radiación

Un total de 82 pacientes con carcinoma de células escamosas de la cabeza y el cuello (SCCHN) se van a aleatorizar en un estudio que se quiere realizar entre enero de 2023 y julio de 2023. Los pacientes reciben la crema de estudio de aplicación tópica o bien el cuidado de la piel "estándar" de los Hospitales donde se realiza el estudio. Todos los pacientes serán tratados con una combinación de radioterapia fraccionada y quimioterapia con base en platino O cetuximab con fines curativos.

El objetivo principal de la crema de estudio es obtener una reducción del número de pacientes que experimenta dermatitis aguda por radiación de grado 3 o 4 (NCI CTCAE versión 4.03) a grado 2, el último día de tratamiento. Como objetivo secundario, obtener una reducción del número de pacientes que experimenta dermatitis aguda por radiación de grado 3 o 4 a grado 0, al mes de finalizar el tratamiento. Se va a evaluar a todos los pacientes periódicamente. Se fotografía la piel irradiada y se clasifican todos los cambios de la dermatitis por radiación. La valoración de la radiodermitis se realizará de modo objetivo mediante u termógrafo. Además, se solicita a los pacientes que cumplimenten cuestionarios acerca de su calidad de vida (QLQ-C30). Estos cuestionarios se responden en las semanas 1, 2 3 y 4 del tratamiento, así como al final de la radioterapia o la quimioterapia.

Para la variable principal de radiodermatitis con CTCAE ≥ grado 2, se realizan evaluaciones según el protocolo (PP), además del enfoque primario de intención de tratar (ITT). En este análisis PP, los pacientes se excluyen de acuerdo con la definición del protocolo o las decisiones de reuniones preanálisis, respectivamente. El estudio se diseña como ensayo aleatorio con una asignación 1:1 a los dos grupos.

El objetivo secundario es estudiar una reducción en el porcentaje de pacientes que experimentan dermatitis por radiación con unos CTCAE máximos de grado 3 o 4 durante el período de tratamiento y en el período de seguimiento de un mes, gracias a la aplicación de la crema de estudio.

#### ANTECEDENTES Y ESTADO ACTUAL DEL TEMA

(Incluyendo bibliografía, máximo 3000 palabras):

La radioterapia (RT) es uno de los principales tratamientos utilizados en oncología para destruir las células tumorales. Es un tratamiento local, con el que únicamente se irradia la zona con células neoplásicas. La radioterapia se puede utilizar como tratamiento principal o como una terapia adyuvante junto con otro tipo de tratamientos como cirugía, quimioterapia, etc.

La piel es la primera barrera que defiende al organismo del exterior y además es un tejido en rápido crecimiento. Aunque en este tipo de tratamiento la piel no es el objetivo primario, acaba siendo blanco de dicha terapia ya que las radiaciones ionizantes tienen necesariamente que atravesarla para alcanzar la zona tumoral.

La dermatitis radioinducida es uno de los efectos secundarios más frecuentes de la radioterapia. Se considera RADIODERMITIS al conjunto de lesiones cutáneas que aparecen tras la exposición de la piel a radiaciones ionizantes, bien con fines terapéuticos o de forma accidental. Existen varias escalas para la clasificación de la severidad de las dermitis inducidas por radiación (RID, de sus



IIS-F-PG-22-02 Edición: 4.2 Página 3 de 18

siglas en inglés, Radiation-induced dermatitis). Una de las más utilizadas es la del National Cancer Institute (USA) (www.nci.org): GRADO 0, sin lesiones; GRADO I, eritema asociado o no a prurito; GRADO II, dermitis seca con prurito más intenso. Eritema moderado, placas con descamación, edema, hiperpigmentación. El daño está confinado a epidermis y dermis; GRADO III, dermitis húmeda, la piel ha perdido su integridad y está húmeda. Descamación confluente mayor a 1,5 cm de diámetro y el daño no está confinado a las capas de la piel. Es más frecuente en las áreas con pliegues como la mama o el cuello. Suele ser dolorosa y más vulnerable a las infecciones. GRADO IV, necrosis cutánea o úlceras. Lesión grave que no es frecuente y su evolución suele ser tórpida.

En la actualidad, no existe un estándar de cuidados ni hay directrices para la prevención y el tratamiento de la dermatitis aguda por radiación. La mayoría de los tratamientos utilizados actualmente son adecuados pero no óptimos en lo que respecta a eficacia y seguridad/tolerancia. Además, la evidencia clínica que respalda su uso es limitada.

El comportamiento específico de un cáncer en particular de cabeza y cuello depende de dónde surge (el sitio primario). Por ejemplo, los cánceres que comienzan en las cuerdas vocales tienen una conducta muy distinta a la de los que surgen en la parte posterior de la lengua, que se encuentra a solamente una pulgada o menos de las cuerdas vocales. El tipo de cáncer más común de cabeza y cuello es el carcinoma de células escamosas, que aparece en las células que revisten el interior de la nariz, la boca y la garganta. El cáncer de células escamosas generalmente se encuentra asociado al consumo de cigarillos o la exposición al virus del papiloma humano (VPH). Otros tipos de cáncer de cabeza y cuello menos comunes son tumores de las glándulas salivales. linfomas y sarcomas. Los métodos de prevención incluyen evitar la exposición a los productos con tabaco y alcohol, como así también vacunar a los niños y a los jóvenes contra el VPH. El cáncer se disemina de cuatro maneras principales. La primera es por extensión directa desde el sitio primario a áreas adyacentes. La segunda es la diseminación a través de los vasos linfáticos hacia los ganglios linfáticos. La tercera es la diseminación a través de los nervios (diseminación perineural) hacia otras áreas de la cabeza y el cuello. La cuarta es la diseminación a través de los vasos sanguíneos a sitios distantes en el cuerpo. En el cáncer de cabeza y cuello, la diseminación a los ganglios linfáticos del cuello es relativamente común. Los ganglios linfáticos que se verán más comúnmente afectados dependerán de la ubicación en la que aparezca el tumor principal. La mayoría de los ganglios linfáticos están ubicados a lo largo de los vasos sanguíneos mayores debajo del músculo esternocleidomastoideo, a cada lado del cuello. El riesgo de diseminación a otras partes del cuerpo por el torrente sanguíneo depende estrechamente de si el cáncer se ha diseminado a los ganglios linfáticos del cuello, cuántos ganglios están afectados, y cuál es su ubicación en el cuello. El riesgo es mayor si hay cáncer en los ganglios linfáticos de la parte inferior del cuello aue que encuentran parte superior (https://www.radiologyinfo.org/es/info/hdneck).

Los cánceres de cabeza y cuello representan casi el 4 % de todos los cánceres en los EE.UU. (<a href="www.cancer.gov">www.cancer.gov</a>) y en la CEE (<a href="www.esmo.org">www.esmo.org</a>). Estos cánceres se presentan con una frecuencia dos veces mayor en hombres que en mujeres. Los cánceres de cabeza y cuello también se diagnostican con mayor frecuencia en personas con más de 50 años de edad que en personas más jóvenes. Utilizando los datos de la incidencia anual de carcinoma de células escamosas de cabeza y cuello (SCCHN), el NCI (USA) estimó que en 2021 hubo 52647 nuevos casos de cáncer de cavidad oral y faringe y 15353 nuevos casos de carcinoma de laringe, lo que ascendió a un total de 68000 casos nuevos de SCCHN. Si el 50% de los pacientes va a ser tratado con radioterapia de haz externo y cabe esperar que el 95% de estos pacientes sufra de dermatitis aguda por radiación,



IIS-F-PG-22-02 Edición: 4.2 Página 4 de 18

lo lógico con esos datos fue esperar que en 2021 hubiera 32300 pacientes que desarrollaron dermatitis aguda por radiación cuando recibieron tratamiento para el SCCHN en los EE.UU.

En este punto es importante destacar que la formulación tópica que proponemos, aunque está dirigida a prevenir las radiodermitis producidas por la radioterapia (y por lo tanto, es de aplicación cutánea), podría perfectamente ser susceptible de aplicación en mucosas y/o tejidos accesibles como por ejemplo la región anal o bucal. Además, dado que las radiodermitis con frecuencia se asocian a dolor, es también de destacar que nuestra formulación es compatible con terapia antiálgica local o general. Existen algunas formulaciones desarrolladas para el tratamiento específico para la radiodermitis, orientadas a la prevención y al tratamiento de las lesiones de la piel inducidas por la radioterapia. Sin embargo, la revisión actualizada sobre los tratamientos disponibles y sus efectos demuestra que su eficacia es muy baja (Lacovelli NA et al. Topical treatment of radiation-induced dermatitis: current issues and potential solutions. Drugs Context. 2020 Jun 12; 9: 2020-4-7). La conclusión de este trabajo de revisión, en el año 2020, es clara: Un producto tópico que contenga componentes seleccionados racionalmente capaces de tratar el dolor, el daño de la piel y los otros síntomas molestos de la dermatitis inducida por radiación, administrado con un vehículo adecuado, asegurando, al mismo tiempo, propiedades quimio-físicas óptimas, podría ser de gran interés en el escenario del tratamiento actual de las dermatitis inducidas por radiación.

La FORMULACION PATENTADA POR NUESTRO GRUPO incide en la protección basándose en varios mecanismos radioprotectores y radiomitigadores de los compuestos en relación a los efectos biológicos de las radiaciones ionizantes. Este avance ha sido recientemente registrado como patente (JM Estrela, E. Obrador y R. Salvador, Universidad de Valencia, UVEG; y A Montoro, Servicio de Protección Radiológica del Hospital Universitario y Politécnico La Fe de Valencia, e investigadora del IIS La Fe): EP21382036 (COMPOSITIONS AND METHODS FOR PREVENTING, AMELIORATING OR REDUCING RADIATION-INDUCED DISEASES). Los 3 principios activos están ampliamente distribuidos a nivel global como cosmeceúticos y nutraceúticos, sin que se hayan reportado efectos negativos.

En octubre de 2022 el grupo consultó a la AEMS para la clasificación de nuestra crema de estudio para futuros estudios en pacientes y la respuesta, por parte del Departamento de Medicamentos de uso humano, Área de ensayos clínicos, fue que Con la información proporcionada la formulación no se considera ni nutracéutico ni producto sanitario. Podrían considerar un cosmético o un medicamento, en función de la finalidad prevista. La finalidad de la crema de estudio para este proyecto propio es que se trata de un preparado que va a estar en contacto con diversas partes superficiales del cuerpo humano, con el fin exclusivo o principal de modificar su aspecto o mantenerlo en buen estado. Las reivindicaciones se circunscribirían estrictamente a una formulación tópica destinada a ayudar a mantener en lo posible la homeostasis fisiológica de la piel.

El grupo de investigación, dentro de los objetivos secundarios del Proyecto AVI que nos ocupa, se propuso el estudio de la Irritación cutánea in vitro: ensayo con modelo de piel humana. Para ello se sub-contrató a la empresa BIONOS, que realizó el estudio de Skin Irritation Test (SIT) utilizando el EpiDerm Skin Model (https://www.mattek.com) y el ensayo de citotoxicidad en queratinocitos (MTT) según las GLP establecidas por la FDA (21 CFR 58) y la OECD, se adjuntan los informes de estos estudios s esta memoria. Además, en estos momentos se está llevando a cabo el estudio en voluntarios sanos para estudiar la cinética de hidratación, cuestionario de autoevaluación subjetiva y efectos antiedad.



IIS-F-PG-22-02 Edición: 4.2 Página 5 de 18

#### HIPÓTESIS DE TRABAJO (máximo 200 palabras):

La protección de la piel en relación a los grados de radiodermitis, en los pacientes con cáncer de cabeza y cuello, sometidos a tratamiento con radioterapia es mayor en los pacientes que han sido tratados con la crema experimental aplicada antes y después de la radioterapia, que en los pacientes tratados con el tratamiento estándar.

Que los pacientes sometidos al tratamiento con la crema de estudio presenten una menor incidencia y grado de radiodermitis, y/o tardanza en el surgimiento de la reacción cutánea a la radiación ionizante, en comparación con los pacientes con cuidado estándar, y todo ello sin diferencias esperadas en las cifras de control tumoral.

#### OBJETIVOS CONCRETOS DE LA INVESTIGACIÓN PROPUESTA (máximo 500 palabras):

#### 1.1. Objetivo principal

El objetivo principal nuestra formulación es estudiar la reducción (en la progresión a dermitis por radiación grave) del número de pacientes que experimentan dermatitis aguda por radiación de grado 3 o 4 a grado 2, el último día de tratamiento. Retraso en aparición de radiodermitis grado 2 respecto al grupo placebo.

#### 1.2. Objetivo secundario

Comparar el porcentaje de pacientes (la incidencia) con radiodermatitis, el grado de toxicidad y el porcentaje de casos con radiodermatitis grado 2 o superior en los pacientes sometidos a los diferentes tratamientos, en la muestra total y estratificada por número de sesiones de radioterapia al mes y al finalizar el tratamiento.

Evaluar y comparar el tiempo para el surgimiento de cada grado de reacción cutánea; identificar la frecuencia y localización de las características específicas de las radiodermatitis.

Estudiar la calidad de vida relacionada con la salud percibida por las pacientes al inicio y al término de la radioterapia. Evaluar y comparar los síntomas locales descritos por los pacientes durante el tratamiento radioterápico y evaluados mediante PREMS-PROMS.

Comparar la temperatura de la zona irradiada mediante un termógrafo durante la radioterapia, en las 4 visitas que realizará el paciente.

#### JUSTIFICACION DEL INTERES DE LA INVESTIGACION PROPUESTA (máximo 1000 palabras):

Aproximadamente el 50 % de todos los pacientes diagnosticados de cáncer en los EE. UU. y Europa recibe tratamiento de radioterapia de haz externo. La dermatitis aguda por radiación se produce aproximadamente en el 95 % de estos pacientes, lo que representa hasta 800 000 pacientes al año en los EE. UU. y 1,7 millones de pacientes al año en Europa.

En la mayoría de los pacientes los efectos de la radioterapia en piel son moderados. Sin embargo, un 20-25% de los pacientes presentan reacciones severas.



IIS-F-PG-22-02 Edición: 4.2 Página 6 de 18

En la actualidad, no existe un estándar de cuidados ni hay directrices para la prevención y el tratamiento de la dermatitis aguda por radiación. La mayoría de los tratamientos utilizados actualmente son adecuados per no óptimos en lo que respecta a eficacia y seguridad/tolerancia. Además, la evidencia clínica que respalda su uso es limitada.



IIS-F-PG-22-02 Edición: 4.2 Página 7 de 18

#### **METODOLOGÍA:**

Por favor, indicar uno por uno todos los puntos que procedan según el tipo de proyecto.

a) <u>Diseño del estudio:</u> (Elementos clave del diseño del estudio que permitan entender el fundamento de este)

El estudio será un estudio clínico con un producto cosmecéutico, randomizado, controlado, paralelo, prospectivo, doble ciego y con dos brazos.

Las cremas (crema experimental (CE) y standard of care (SC)) se distribuirán aleatoriamente entre los pacientes, de forma que un 50% reciban CE y el otro 50% SC. Cada tubo tendrá un nº cuyo contenido no conocerán ni los evaluadores ni los pacientes.

En un periodo comprendido entre enero de 2023 y junio de 2023, los servicios de oncología radioterápica de los Hospitales La Fe y Clínico de Valencia, realizarán un estudio a 82 pacientes con SCCHN. Que serán sometidos a radioterapia de haz externo con o sin quimioterapia concomitante.

El tratamiento radioterápico emplea técnicas de intensidad modulada del haz de radiación (IMRT o VMAT) guiadas por la imagen (IGRT) que ofrecen una muy alta precisión en la administración diaria del tratamiento, mejorando la tolerancia de los tejidos sanos y la calidad de vida de los pacientes.

Los pacientes serán distribuidos en dos grupos:

Grupo A (intervención, CE): este grupo recibirá la aplicación tópica de la crema de estudio.

Grupo B (control, SC): a este grupo se le aplicará el standard care

#### Tratamiento de estudio

Los pacientes recibirán la instrucción de aplicar la crema en el área a ser irradiada, 2 veces al día, cada ocho horas aproximadamente (mañana, tarde y noche); siempre, después de la sesión de radioterapia y comenzando dos días antes al día de inicio de la radioterapia, para evitar la aplicación de la crema justo antes de la sesión.

#### Tratamiento control

El estándar de tratamiento para la dermatitis por radiación en los Servicios de Oncología Radioterápica, es utilizar un *standard care*. En el brazo de control del estudio, a los pacientes se les proveerá de botes de crema aleatorizados con el SC.

También recibirán instrucciones para seguir el protocolo de prevención de radiodermatitis con cuidados estandarizados consensuados por los dos servicios de oncología radioterapia de los dos Hospitales que participan. Protocolo de prevención de radiodermatitis:

El protocolo estándar incluye instrucciones generales para prevenir que el área de la piel irradiada sea afectada que se proporcionan a todos los pacientes tratados con radioterapia y en este caso consensuado para los dos Hospitales.

Los participantes serán distribuidos aleatoriamente en dos grupos. La randomización se hará en bloques y estará estratificada por número de sesiones de radioterapia, utilizando el programa estadístico R 4.0.2(R Core Team, 2022; Viena, Austria).

En el caso del presente estudio, el tratamiento consistirá en x sesiones, con entrega de dosis fraccionada en días hábiles (excluyendo fines de semana). Los pacientes recibirán 3 volúmenes diferentes de esquemas de irradiación, una dosis máxima de 70 Gy (2Gy/ fracción/ día, otro grupo de pacientes con un esquema de 63



IIS-F-PG-22-02 Edición: 4.2 Página 8 de 18

Gy (1,8 Gy/ fracción/día) y el tercer grupo de pacientes, con una dosis total de 54-56 Gy (1,6 Gy/ fracción/día). Antes de iniciar el tratamiento, las pacientes tendrán una consulta con enfermería, donde se explicarán las orientaciones generales y de prevención de los efectos adversos.

**b)** <u>Contexto:</u> (descripción del marco, los lugares y las fechas relevantes, incluyendo fechas de reclutamiento, exposición, seguimiento y recogida de datos)

Los pacientes van a comenzar la radioterapia fraccionada estándar pudiendo ser concomitante con la quimioterapia y ésta podría ser platino o cetuximab y con una duración del tratamiento de entre 6 y 8 semanas.

#### Fechas relevantes:

Cada paciente participará en el estudio durante aproximadamente 3 meses, que incluirá una semana Para el período de selección, 5 a 8 semanas de tratamiento y asistencia a la clínica de seguimiento. Se realizarán cuatro visitas clínicas, desde una semana antes del inicio de la radioterapia, para evaluar a cada paciente (primera visita al hospital), hasta 2 semanas después del final de la radioterapia (cuarta visita al hospital).

La segunda visita clínica de seguimiento y la evaluación será a las 4 semanas después del inicio del tratamiento con radiación. La tercera visita clínica de seguimiento y evaluación será al final del tratamiento con radiación. La cuarta y última visita de seguimiento y evaluación de la clínica será 2 semanas después del final del tratamiento con radiación.

La duración total del estudio será de aproximadamente de 12 semanas para pacientes con SCCHN.

En cada visita a la consulta clínica, se recopilará información del paciente relacionada con cambios en la piel debidos a la radiación, examen físico y evaluación de la calidad de vida.

El análisis de datos de los pacientes y la clasificación de la dermatitis por radiación, si se produce, se realizará en 3 de las visitas clínicas de seguimiento, la segunda, tercera y cuarta (última) (Tabla 2).

| Categoría | Información |
|---|---|
| | Tipo histológico |
| Tumor | Estadio (tumor, nodo, metástasis) |
| | Localización |
| | Edad |
| | Hábito tabáquico (0=No, 1=Hasta 10 cig/dia; 2= +10 cig/años) |
| Paciente | Período de exposición al tabaco (años) |
| | Alcohol |
| | Etnia |
| | Peso |
| | Comorbilidad (por ejemplo, diabetes, enfermedades relacionadas con el colágeno, hipertension, inflamac |
| | _ |
| | Intención de tratamiento (radical o adyuvante) |
| Tratamiento | Uso de quimioterapia |
| | Tipo de quimioterapia (cisplatino y cetuximab) |



IIS-F-PG-22-02 Edición: 4.2 Página 9 de 18

| | Uso de cirugía |
|---|---|
| | Complicaciones postoperacionales |
| | Medicación concurrente (como estatinas) |
| | Dosis total de radiación |
| Física | Dosis por fracción |
| 1 13100 | Tiempo total de tratamiento |
| | Dosis a piel |
| | Datos pretratamiento |
| | Datos muestra recogida al final del tratamiento |
| Toxicidad | Datos muestra recogida 6 meses después |
| Toxicidad | Datos muestra anual |
| | Clasificación de la toxicidad por el criterio de la RTOG por órgano/tejido |
| | Toxicidad valorada por el especialista |

| | Primera visita<br>clínica: 7 días<br>después de<br>empezar QRT | Segunda visita clínica: 3-4 semanas después de empezar QRT | Tercera visita<br>clínica: al<br>finalizar QRT | Cuarta visita clínica: 2 semanas después de acabar QRT |
|---|---|---|---|---|
| Evaluación del | | | | |
| paciente | | | | |
| Firma del | | | | |
| consentimiento | | | | |
| informado | | | | |
| Datos | | | | |
| demográficos | | | | |
| (edad, sexo, tipo | | | | |
| de tumor, grado, estadío | | | | |
| Historia médica y | | | | |
| examen físico | | | | |
| Clasificación de la | | | | |
| radiodermitis, | | | | |
| termografía (y | | | | |
| fotografías) | | | | |
| Completar | | | | |
| cuestionarios | | | | |
| calidad de vida | | | | |

Tabla 2. Calendario del estudio y visitas clínicas de seguimiento del paciente antes, durante y después de la QRT

Previo a estas sesiones, donde se valorarán una serie de parámetros clínicos de rutina en estos pacientes en este servicio, habrá una primera visita donde se explicará al paciente el proyecto de investigación, se le entregará la hoja de información y el consentimiento informado.



IIS-F-PG-22-02 Edición: 4.2 Página 10 de 18

Tabla 3: Se presenta a continuación cada objetivo de este estudio y en qué momento se evalúa:

| Objetivos | | 2ª visita: 3-4 s. | | |
|---|---|---|---|---|
| | QRT | tras QRT | finalizar QRT | tras fin QRT |
| Principal | | | | |
| Obtener una reducción grado radiodermitis grado 3-4 a 2 | | | | X |
| Secundarios: | | | | |
| Porcentaje de pacientes con radiodermitis | | | | Х |
| Porcentaje de pacientes con grado de toxicidad 3-4 | | | | Х |
| Porcentaje radiodermitis en la muestra total | | | | Х |
| Porcentaje radiodermitis en la muestra estratificada | | | | Х |
| Frecuencia y localización de las características específicas radiodermitis | X | X | X | X |
| Valoración objetiva de la radiodermitis mediante termógrafo | X | X | X | X |

# c) Participantes

#### - Criterios de eligibilidad

Pacientes mayores de edad que van a ser tratados con radioterapia externa de carcinoma de células escamosas de cabeza y cuello que acuden al Servicio de Oncología Radioterápica del Hospital Universitario y Politécnico la Fe de Valencia.

#### Criterios de inclusión

Se van a reclutar pacientes con SCCHN localizado (no metastásico) confirmado histológicamente. Los pacientes tienen 18 años o más, con ECOG (Eastern Cooperative Oncology Grupo) Estado funcional de rendimiento de 0 a 2, una esperanza de vida de 6 meses o más, y con el consentimiento informado firmado. Piel íntegra al inicio de la radioterapia.

#### - Criterios de exclusión

Los pacientes serán excluidos si tienen metástasis a distancia, radioterapia previa para SCCHN, participación en curso en cualquier otro estudio o ensayo clínico.

Las pacientes que estaban embarazadas o en periodo de lactancia serán excluidas del estudio, al igual que aquellos con hipersensibilidad conocida a cualquiera de los componentes de la crema de estudio.

Los pacientes con cáncer previo o concurrente dentro de los 5 años de comienzo del estudio y cualquier otra condición social o médica que pueda afectar la participación en o evaluación del estudio serán excluidos.

Tener antecedentes de enfermedad del colágeno, como lupus eritematoso sistémico y/o esclerodermia.

Presentar afecciones dermatológicas, como psoriasis, pénfigo bulloso o epidermólisis ampollosa o bullosa.



IIS-F-PG-22-02 Edición: 4.2 Página 11 de 18

Tener alteraciones inflamatorias visibles en la piel del área a ser irradiada

Criterios de retirada de los sujetos

Los sujetos pueden retirar su consentimiento para su participación en cualquier momento sin perjuicio. Adicionalmente, el investigador puede retirar a un sujeto si, según la opinión clínica del investigador, está en el mejor interés del sujeto o si el sujeto no puede cumplir con los requisitos del protocolo.

El promotor puede interrumpir el protocolo en cualquier momento. Los motivos para detener el estudio pueden incluir, pero no se limitan a, los siguientes:

- Incidencia inaceptable de acontecimientos adversos
- Inclusión inadecuada de sujetos
- Recogida de datos inadecuada o imprecisa

En caso de que el paciente presente radiodermatitis de grado 1 o 2, el protocolo del estudio se mantendrá inalterado con la continuación de la aplicación de la crema, ya que el tratamiento estándar de estas lesiones es la aplicación de hidratantes tópicos, función ya desempeñada por la crema estudiada.

En caso de que el paciente presente radiodermatitis de grado 3 o 4, la radioterapia y la aplicación de la crema podrán ser suspendidas por el médico radioterapeuta hasta que la lesión de piel mejore; el tratamiento tópico de las lesiones corresponderá a sus características, conforme con el protocolo institucional. El paciente deberá continuar aplicando la crema en las regiones irradiadas no afectadas por la lesión.

- Métodos de seguimiento

La clasificación del grado de dermatitis por radiación que se va a utilizar en el seguimiento y valoración de la radiodermitis serán los sistemas de clasificación visual del Instituto Nacional del Cáncer (NCI), los Criterios de Toxicidad Comunes para Eventos Adversos (CTCAE)

## d) Variables

Pacientes mayores de edad de ambos sexos con tumores de cabeza y cuello.

Las variables del proyecto se detallan a continuación:

#### VARIABLES DEMOGRÁFICAS

SIP

Fecha de nacimiento: día/mes/año.

Sexo: Hombre o mujer. Antecedentes personales.

Tratamiento farmacológico habitual.

#### **VARIABLES CLÍNICAS**

DIAGNÓSTICO

Fecha Biopsia: mes/año.



IIS-F-PG-22-02 Edición: 4.2 Página 12 de 18

```
Histología:
       Carcinoma epidermoide
       Carcinoma adenoide quístico
               Indiferenciado
       Otra:
       Localización tumor primario:
       Cavidad oral:
               Labio
               Suelo de boca
               Encia
               Lengua
       Orofaringe
               Base de lengua
               Fosa amigdalina
               Trígono retromolar
               Pared posterior faríngea
       Glándula salivar
               Submaxilar
               Parótida
       Estadío: I, II, III o IV.
TRATAMIENTO
       CIRUGIA: Si o No.
       Fecha de cirugía: día/mes/año.
       QUIMIOTERAPIA: Si o No.
       Fecha de inicio de QT: día/mes/año.
       Fecha fin QT: día/mes/año.
       Tipo de QT:
       Neoadyuvante
       Adyuvante
               Radical
       Citostático:
       DCF
       CDDP 100
       CTX
       CDDP 40
               DCF seguido de CDDP 100
               DCF seguido de CDDP 40
               DCF seguido de CTX
               Otro
       RADIOTERAPIA
       Fecha de inicio de RT: día/mes/año.
       Fecha de fin RT: día/mes/año.
       Tipo de RT:
       Radical
       Adyuvante
       Campo de RT:
       Cuello unilateral derecho.
       Cuello unilateral izquierdo.
       Cuello bilateral.
       Dosis media alcanzada en piel de cuello:
       Lado derecho:
       Lado izquierdo:
       Dosis máxima alcanzada en piel de cuello.
       Lado derecho:
```



IIS-F-PG-22-02 Edición: 4.2 Página 13 de 18

Lado izquierdo:

#### VARIABLES ESPECIFICAS

(Para recoger la toxicidad cutánea propongo seguir los criterios de CTCAE v. 5.0) TOXICIDAD CUTÁNEA AGUDA (CTCAe V.5):

| | | Skin and subcutaneous tissue | disorders | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Skin atrophy | Covering <10% BSA; | Covering 10 - 30% BSA; | Covering >30% BSA; | - | - |
| | associated with | associated with striae or | associated with ulceration | | |
| | telangiectasias or changes in | adnexal structure loss | | | |
| | skin color | 1 | | | |
| Definition: A disorder charact | terized by the degeneration and thinn | ing of the epidermis and dermis. | | | |
| Navigational Note: - | | | | | |
| Skin hyperpigmentation | Hyperpigmentation covering | Hyperpigmentation covering | - | - | - |
| | <10% BSA; no psychosocial | >10% BSA; associated | | | |
| | impact | psychosocial impact | | | |
| Definition: A disorder charact | terized by darkening of the skin due to | excessive melanin deposition. | | | |
| Navigational Note: - | | | | | |
| Skin hypopigmentation | Hypopigmentation or | Hypopigmentation or | - | - | - |
| | depigmentation covering | depigmentation covering | | | |
| | <10% BSA; no psychosocial | >10% BSA; associated | | | |
| | impact | psychosocial impact | | | |
| Definition: A disorder charact | terized by loss of skin pigment (e.g., vi | tiligo). | | | |
| Navigational Note: - | | | | | |
| Skin induration | Mild induration, able to move | Moderate induration, able to | Severe induration; unable to | Generalized; associated with | Death |
| | skin parallel to plane (sliding) | slide skin, unable to pinch | slide or pinch skin; limiting | signs or symptoms of impaired | |
| | and perpendicular to skin | skin; limiting instrumental ADL | joint or orifice movement | breathing or feeding | |
| | (pinching up) | | (e.g., mouth, anus); limiting | | |
| | | | self care ADL | | |
| Definition: A disorder charact | terized by an area of hardness in the s | kin. | | | |
| Navigational Note: - | | | | | |
| Skin ulceration | Combined area of ulcers <1 | Combined area of ulcers 1 - 2 | Combined area of ulcers >2 | Any size ulcer with extensive | Death |
| | cm; nonblanchable erythema | cm; partial thickness skin loss | cm; full-thickness skin loss | destruction, tissue necrosis, or | |
| | of intact skin with associated | involving skin or | involving damage to or | damage to muscle, bone, or | |
| | warmth or edema | subcutaneous fat | necrosis of subcutaneous | supporting structures with or | |
| | | | tissue that may extend down | without full thickness skin loss | |
| | | | to fascia | | |
| Definition: A disorder charact | terized by a circumscribed, erosive les | ion on the skin. | | | |

Clasificación CTCAE de la dermatitis por radiación. El grado de dermatitis por radiación se evalúa utilizando el CTCAE del Instituto Nacional del Cáncer clasificación (V.4.03).8-10 La documentación fotográfica de las lesiones cutáneas se realizó.

Grados de lesión: Eritema, Hidratación, Pigmentación, Elasticidad de la piel.

A continuación, se describe la apariencia de la piel para cada grado:

Dermatitis por radiación leve, grado 1 de CTCAE: el inicio se produce entre días y semanas después de comenzar la terapia, pero los síntomas pueden desaparecer en un mes. La piel muestra un eritema leve que palidece con la compresión o "descamación seca". Se puede observar prurito y caída del cabello.

Dermatitis por radiación moderada, CTCAE grado 2: Esto puede ser más grave 1 a 2 semanas después el final del tratamiento. La piel muestra un intenso edema y eritema que es doloroso, y esto puede progresar a la pérdida de la epidermis y a la "descamación húmeda" que incluye exudados fibrinosos y ampollas.

Dermatitis por radiación grave, grado 3 de CTCAE: esta forma de dermatitis incluye dermatitis húmeda confluente descamación que puede progresar a necrosis y ulceración de la piel en todo el espesor. El dolor puede ser bastante severo.

Dermatitis por radiación grave, grado 4 de CTCAE: Esta es una forma rara de dermatitis, que ocurre en menos del 5% de los pacientes, e incluye necrosis y ulceración de la piel de espesor total. Puede requieren la interrupción de la radioterapia y el tratamiento con desbridamiento quirúrgico, injerto de piel de espesor total o cirugía reconstructiva.



IIS-F-PG-22-02 Edición: 4.2 Página 14 de 18

#### Cuestionarios de calidad de vida

Todos los pacientes reciben cuestionarios EORTC QOL, (QLQ) C30 (30 preguntas) (versión 3), (QLQ) Cabeza y Cuello (H&N) C30 (65 preguntas) (versión 3). Los cuestionarios se completan en cada visita al Hospital en el seguimiento desde el día de la evaluación inicial (primera visita a la consulta clínica) hasta 2 semanas postratamiento (cuarta visita a la consulta clínica).

## Termógrafo

Uso de las características texturales y basadas en la temperatura como biomarcadores de imágenes para la dermatitis inducida por radiación.

Uso del termógrafo (es decir, termorradiomia) para desarrollar una herramienta predictiva para la toxicidad de la piel inducida por radiación en los primeros intervalos de tiempo del tratamiento. Se medirán las características térmicas de la piel irradiada en pacientes con cáncer cabeza y cuello. La toxicidad de la piel inducida por la radiación está asociada con un aumento en la temperatura de la superficie de la piel y cambios en los parámetros termorradiómicos.

## e) <u>Tamaño muestral</u> (explicar además cómo se determinó)

Aceptando un riesgo alfa de 0.05 y un riesgo beta de 0.2 en un contraste bilateral, se precisan 41 sujetos en el primer grupo y 41 en el segundo para detectar como estadísticamente significativa la diferencia entre dos proporciones, que para el grupo 1 se espera sea de 0.1 y el grupo 2 de 0.35. Se ha utilizado la aproximación del ARCOSENO.

f) <u>Métodos estadísticos</u> (en el protocolo de investigación los investigadores deben determinar por anticipado al menos los análisis para los objetivos primarios del estudio)

Las variables cualitativas serán descritas mediante frecuencias y porcentajes mientras que las variables cuantitivas mediante media y su desviación estándar. Se comprobará la normalidad de las variables continuas mediante el test de Shapiro-Wilks y en caso de no confirmarse su distribución normal serán descritas mediante mediana y rango intercuartílico.

El objetivo principal de este estudio será analizado mediante un test de proporciones. Los tres primeros objetivos secundarios serán evaluados en función al tipo de variable estudiada. En caso de variables cuantitativas se realizará comparación de medias mediante T-Student en caso de existir normalidad o el test de Mann-Whitney en caso contrario. Para las variables cualitativas se realizará comparación de porcentajes entre grupos por medio del test exacto de Fisher o mediante test de ji-cuadrado según convenga. El último de los objetivos secundarios será estudiado mediante un análisis de varianza con medidas repetidas en caso de aceptarse la normalidad de los residuos y el test de Friedman en caso contrario.

La aleatorización de los pacientes será simple al azar. El proceso para ello será mediante el software estadístico R (R Core Team, 2022) utilizando el paquete randomizeR (Uschner et al. 2018). Uschner D, Schindler D, Hilgers R, Heussen N (2018). "randomizeR:An R Package for the



IIS-F-PG-22-02 Edición: 4.2 Página 15 de 18

| Assessment and Implementation of Randomizationin Clinical Trials." _Journal of Statistical Software_, *85*(8), 1-22. doi:10.18637/jss.v085.i08 <a href="https://doi.org/10.18637/jss.v085.i08">https://doi.org/10.18637/jss.v085.i08</a> >. |
|---|
| R Core Team (2022). R: A language and environment for statistical computing. R Foundation for Statistical Computing, Vienna, Austria. URL <a href="https://www.R-project.org/">https://www.R-project.org/</a> . |
| Para homogeneizar la forma de administración de las cremas de estudio hay que resaltar que todos los pacientes pasarán por una consulta de enfermería donde se les explicará cómo administrarse las cremas. |
| g) Calendario y plan de trabajo (con fecha de inicio y fin de proyecto) |
| Enero 2023 hasta julio 2023 |
| Enero 2023 hasta julio 2023 |



IIS-F-PG-22-02 Edición: 4.2 Página 16 de 18

#### TÍTULO DEL PROYECTO DE INVESTIGACIÓN:

Desarrollo de una crema protectora frente a las radiodermitis causadas por la radioterapia.

## **MEMORIA ECONÓMICA**

1. Coste que la realización del proyecto puede suponer:

Desglose del presupuesto previsto para el proyecto de investigación, indicando la cuantía de dinero a gastar por partida de gasto y anualidad (máximo 5 años).

| PARTIDAS | | | | |
|---|---|---|---|---|
| | Año 1 | Año 2 | Año 3 | Total |
| Gastos de personal | 10468,44 | | | 10468,44 |
| Material fungible | 28500 | 58600 | | 87100 |
| Material inventariable<br>/equipamiento | 6000 | 7124 | | 13124 |
| Subcontratación de<br>servicios | 7100 | 134350 | 115520 | 256700 |
| Registro propiedad | | 12000 | 32000 | 44000 |
| Auditoria | 800 | 800 | 800 | 2400 |
| Cargos internos<br>(Plataformas CientfTec. IIS) | | | | |
| Formación y otros gastos<br>(congresos, viajes y<br>desplazamientos, dietas y<br>manutención) | | | | |
| Publicaciones y revistas<br>científicas | | | 3000 | |
| COSTE TOTAL | 52868,44 | 223342,44 | 151050 | 427260,88 |

A continuación se explica el destino de las diferentes partidas:

En concreto para el este estudio en pacientes es el montante de 157.624 euros, repartido en dos Hospitales el específico para el estudio en pacientes. En relación a este montante, la cantidad de dinero:

# Estudio en pacientes:

Hospital la Fe, estudio en pacientes año 2022: 32.625 € y para el año 2023: 32.625 € Hospital Clínico, estudio en pacientes año 2022: 32.625 € y para el año 2023: 32.625 € Total para los dos hospitales y los dos años: 130.500 €\*

\*Esta cantidad incluye pago a clínicos por estudio de cada paciente, análisis estadístico INCLIVA, pago por el apoyo al servicio de Coordinación de ensayos del IISLAFE y a otros departamentos implicados del IISLAFE.

## El seguro de pacientes:

Hospital la Fe, estudio en pacientes año 2022: 5000 € y para el año 2023: 5000 € Hospital Clínico, estudio en pacientes año 2022: 5000 € y para el año 2023: 5000 €



IIS-F-PG-22-02 Edición: 4.2 Página 17 de 18

Total para los dos hospitales y los dos años: 20.000 €

# Equipamiento:

Termógrafo para Hospital La Fe: 7.124 €

Del montante global del proyecto concedido, de 427.260,88 €, para el estudio en los pacientes para dos Hospitales es de **157.624** €

# 2. Financiación prevista para el proyecto:

## 2.1 DISPONIBLE ACTUAL:

| Proyecto/s de partida indicar referencia IIS La Fe | Cuantía de dinero a traspasar |
|---|---|
| 00700405-LÍNEA DE INVESTIGACIÓN<br>DESARROLLO Y TRANSFERENCIA DE | 85250 euros |
| CONTRAMEDIDAS MÉDICAS | 30200 Gui GG |

| PARTIDAS | | | | |
|---|---|---|---|---|
| PARTIDAS | Año 1 | Año 2 | Año 3 | Total |
| Gastos de personal | | | | |
| Material fungible | | | | |
| Material inventariable /equipamiento | | | | |
| Subcontratación de servicios | | 42625 | 42625 | 42625 |
| Cargos internos<br>(Plataformas CientfTec. IIS) | | | | |
| Formación y otros gastos<br>(congresos, viajes y<br>desplazamientos, dietas y<br>manutención) | | | | |
| Publicaciones y revistas científicas | | | | |
| TRASPASO TOTAL | | 42625 | 42625 | 85250 |

## 2.2 PREVISIÓN FUTURA:

2.2.1 Fuente de financiación: FONDOS PROPIOS



IIS-F-PG-22-02 Edición: 4.2 Página 18 de 18

| | PERIODO DE EJECUCIÓN | | | | | |
|---|---|---|---|---|---|---|
| Donaciones / Convenios² / Patrocinios/ Prestación de servicios / Traspasos EECC/Bolsas | Año 1 | Año 2 | Año 3 | Año 4 | Año 5 | Total |
| Total | | | | | | |

2.2.2 Otras fuentes de financiación (especificar):

 $<sup>^2</sup>$  Tabla 2.2.1 Fuentes de financiación: Fondos propios: indicar la entidad financiadora en los casos que corresponda.